CLINICAL TRIAL: NCT00582439
Title: The Use of the Reamer-Irrigator-Aspirator (RIA) to Harvest Bone Graft for Treatment of Non-unions and Fractures
Brief Title: The Use of RIA to Harvest Bone Graft for Treatment of Non-unions and Fractures
Acronym: RIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Synthes Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F061229004
Record Dates: First submitted 2007-12-20; First posted 2007-12-28 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Orthopaedic Trauma Fractures and Non-unions
Keywords: Orthopaedic Trauma Fractures; Orthopaedic Trauma Non-unions; Reamer-Irrigator-Aspirator (RIA); Bone Graft
MeSH Terms: interventions — Radioimmunoassay

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Repair of Orthopaedic Trauma Fractures and Non-Unions
  Interventions: Device: Reamer-Irrigator-Aspirator (RIA)

INTERVENTIONS:
Device: Reamer-Irrigator-Aspirator (RIA) — Patients must already be scheduled for bone grafting of a fracture or nonunion with harvest of autologous graft material from their femur using the RIA system. The reaming procedure will be conducted using the trochanteric entry portal through the tip of the greater trochanter.
  Other Names: Reamer-Irrigator-Aspirator (RIA), Synthes, Inc.

SUMMARY:
This study is to determine the composition of bone graft harvested using the RIA system in 16 orthopaedic trauma patients between age 19 and 65 who have sustained a fracture or non-union requiring bone grafting. The patients will be followed to assess clinical outcomes and associated pain.

DETAILED DESCRIPTION:
Early clinical use has suggested that bone graft obtained from the human femur using the RIA system is available in large quantities, may be associated with less pain when compared to conventional methods of autograft harvest, and may provide bioactive substances in addition to bone that aid in the healing process.

All patients enrolling in this study will be scheduled for bone grafting of their fracture or nonunion using the RIA system, irregardless of their participation in the study. There is pain associated with the harvest of the bone, but it will be the same whether the patient is enrolled in the study or not.

A total of sixteen patients will be enrolled in this study, eight will have large (2.8 - 5.6 mm) Beta-Tricalcium Phosphate (ChronOS) granules in the second filter, eight will have medium (1.4 - 2.8 mm) Beta-Tricalcium Phosphate (ChronOS)granules. All patients will be enrolled after obtaining informed consent. In order to be eligible for the study, the patients must already be scheduled for bone grafting of a fracture or nonunion with harvest of autologous graft material from their femur using the RIA system. The reaming procedure will be conducted using the trochanteric entry portal through the tip of the greater trochanter. The reamer size will be determined using fluoroscopy to measure the medullary canal at the isthmus of the femur. All bone graft harvest will be obtained using a single pass reaming over a guide wire placed centrally in the distal femur. Two 750 micrometer filters will be placed in series at the suction end of the RIA. The first filter will collect the bone, and the second filter will be filled with Beta-Tricalcium Phosphate. Three samples (< 1 cc) of the bone will be collected from the first filter. The first sample will be from the top of the filter, the second sample will be obtained halfway down the filter, and the final sample will be obtained from the bottom of the filter. Similarly, three samples of Beta-Tricalcium Phosphate will be obtained from the second filter. Each of these samples will also be less than 1 cc of material. The first sample will be from the top layer, the second sample will be from the middle of the Beta-Tricalcium Phosphate layer, and the final sample will be from the bottom of the filter. The middle of each filter layer will be determined by measuring the filter sample with a ruler and dividing by two. Each of these samples will be stored in dry ice and transported to the Department of Surgery laboratories run by Dr. Irshad Chaudry for processing as described below. We will also obtain a single sample of the fluid effluent that is normally discarded as part of the procedure. That sample will be analyzed for the same proteins and factors described below.

All patients will undergo a needle biopsy of their ipsilateral iliac crest while under general anesthesia for their surgical procedure. The bone biopsy will be taken through the surgical incision used for placing the reamer irrigator aspirator in most cases. If a patient requires only a small incision for placing the reamer, which precludes needle biopsy through the surgical incision, then the needle biopsy will occur through a small (< 1 cm) incision directly over the iliac crest. The iliac crest biopsy will also be immediately placed on dry ice and transported to the Department of Surgery laboratories of Dr. Chaudry for evaluation. After the samples have been obtained, the scheduled surgical procedure will be completed.

ELIGIBILITY:
Inclusion Criteria:

* patient must have a fracture or non-union requiring bone grafting
* adult patient between ages 19 and 65

Exclusion Criteria:

* primary bone tumors or known metastatic disease involving the bone
* patients with osteomyelitis in the femur that will be used to harvest bone graft
* patients unable or unwilling to give informed consent

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-01; Primary Completion 2007-05 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Treatment of Nonunions and Fractures with Bone Graft | Recruitment:: 1 day; Surgery: 1 day; Follow-up: 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David A Volgas, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Orthopaedic Trauma, Birmingham, Alabama, United States

REFERENCES:
- [Background] Hammer TO, Wieling R, Green JM, Sudkamp NP, Schneider E, Muller CA. Effect of re-implanted particles from intramedullary reaming on mechanical properties and callus formation. A laboratory study. J Bone Joint Surg Br. 2007 Nov;89(11):1534-8. doi: 10.1302/0301-620X.89B11.18994. PMID 17998197